CLINICAL TRIAL: NCT07023523
Title: Self-regulation of Real-time fMRI Brain Activity in Chronic Pain: A Potential Neurobiological Mechanism of Cognitive Behavioral Therapy
Brief Title: Self-regulation of Real-time fMRI Brain Activity in Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Jeungchan Lee, Assistant Professor, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: R21AR084246 (NIH); R21AR084246 (NIH)
Record Dates: First submitted 2025-06-03; First posted 2025-06-17 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study personnel collecting, entering, and analyzing data are blind to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): 8 individual weekly visits with a psychologist for pain-related CBT.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Disease Education (Active Comparator): 8 individual weekly visits with a psychologist for fibromyalgia education (this is an active comparator arm, matched for provider contact).
  Interventions: Behavioral: Disease Education

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Practicing certain cognitive and behavioral pain self-management strategies such as relaxation and changing negative thoughts about pain.
  Arms: Cognitive Behavioral Therapy
Behavioral: Disease Education — Providing information about fibromyalgia, including its potential causes and management approaches.
  Arms: Disease Education

SUMMARY:
This study aims to explore the usefulness of self-regulation of brain activity in patients with fibromyalgia. Patients will use real-time functional magnetic resonance imaging (fMRI) neurofeedback to observe and regulate their own brain activity while applying mental strategies to reduce fibromyalgia pain. The study consists of 2 magnetic resonance imaging (MRI) visits that involve brain neuroimaging for fMRI neurofeedback tasks, as well as 8 weekly intervention sessions with a pain psychologist. Patients will be randomized to either Cognitive Behavioral Therapy (CBT) or Fibromyalgia Education groups.

DETAILED DESCRIPTION:
Pain catastrophizing-a negative cognitive and emotional process that involves helplessness, rumination, and magnification of pain complaints-is the most consistent psychosocial factor predicting deleterious outcomes in chronic musculoskeletal pain, including fibromyalgia. We will use real-time functional magnetic resonance imaging (fMRI) neurofeedback as a research probe to elucidate the neurological mechanisms underlying self-regulation of pain catastrophizing in individuals with fibromyalgia.

Investigators will recruit patients diagnosed with fibromyalgia. In the baseline magnetic resonance imaging (MRI) visit, participants will complete a fMRI neurofeedback session inside an MRI scanner. Prior to entering the scanner, participants will complete several questionnaires and discuss with the research team the self-regulation strategies they plan to use during the neurofeedback task to modulate fibromyalgia pain. For the neurofeedback, participants will be presented with a visual representation of their brain activity performance so that they can maintain or update their strategy throughout the run. As part of the baseline visit, investigators will also apply moderate pressure pain to the patient's leg in the scanner to see how their brain responds to the experimental pain stimulation.

After the baseline visit, participants will be randomly assigned into the Cognitive Behavioral Therapy (CBT) or Fibromyalgia Education groups, and they will then attend 8 weekly intervention sessions with a pain psychologist. During the post-intervention MRI visit, participants will complete the same questionnaires and tasks performed at the baseline visit to assess changes in neural mechanisms underlying the self-regulation of fibromyalgia pain and the experience of experimental pain. All outcome measures will be assessed at both baseline and post-intervention visits.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65
2. Meet the Wolfe et al 2011 research criteria for fibromyalgia for at least one year
3. On stable doses of medication prior to entering the study and agree not to change medications or dosages (or CAM treatments) during the trial
4. Baseline pain intensity of at least 4/10 on average and pain report for at least 50% of days
5. Able to provide written consent and fluent in English

Exclusion Criteria:

1. Comorbid acute pain condition
2. Comorbid chronic pain condition that is rated by the subject as more painful than fibromyalgia
3. Stimulant medications for the fatigue associated with sleep apnea or shift work (e.g., modafinil),
4. Pregnant or nursing
5. Any psychiatric disorder involving a history of psychosis (e. g schizophrenia, severe personality disorders)
6. History of anxiety disorders or significant anxiety symptoms interfering with fMRI procedures (e.g., panic)
7. Contraindication to MRI (e.g., implanted ferrous metal)
8. History of significant head injury (e.g., with substantial loss of consciousness)
9. Psychiatric hospitalization in the past 6 months
10. Other contraindications to MRI
11. Participating in other therapeutic trials
12. Active suicidal ideation
13. Documented peripheral neuropathy of known cause (e.g diabetic neuropathy, chemotherapy-induced neuropathy, guillain-barre)
14. Routine or daily use of narcotics or substances of abuse
15. Autoimmune or inflammatory disease (RA, SLE, IBD) that causes pain
16. Lower Limb Vascular Surgery or Current Lower Limb Vascular Dysfunction
17. Any impairment, activity or situation that in the judgment of the Study Coordinator or Principal Investigator that would prevent satisfactory completion of the study protocol. This includes unreliable, or inconsistent pain scores as deemed by the principal investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Changes in brain activity in pain-associated regions such as vPCC/RSC | Brain activity data will be collected at baseline and at post-treatment, spanning approximately 4 months.
  Changes in brain activity in pain-associated regions such as vPCC (ventral posterior cingulate cortex)/RSC (retrosplenial cortex), quantified as z-scores, during the self-regulation period of the MRI scan.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale (PCS) | PCS will be assessed at baseline and at post-treatment, spanning approximately 4 months.
  Pain catastrophizing will be assessed with the Pain Catastrophizing Scale (PCS).
  Pain Catastrophizing Scale (PCS) is a validated survey instrument that assesses the extent of catastrophizing thinking related to pain. Pain catastrophizing is assessed on a scale from 0 to 52, with higher scores indicating a higher levels of catastrophizing.
Brief Pain Inventory (BPI) | BPI will be assessed at baseline and at post-treatment, spanning approximately 4 months.
  Brief Pain Inventory (BPI) is a validated questionnaire designed to assess the severity and interference of pain experienced. Pain severity is assessed on a scale from 0 (no pain) to 10 (severe pain). Pain interference is assessed on a scale from 0 (no interference) to 10 (severe interference).

OTHER OUTCOMES:
Self-regulation performance | Self-regulation performance will be assessed at baseline and at post-treatment, spanning approximately 4 months.
  During each real-time fMRI self-regulation trial, patients will receive visual feedback of their modulated brain activity, and neurofeedback performance will be measured by their ability to successfully modulate the visual feedback indicator (i.e., increasing/decreasing it as instructed). Changes in performance scores between baseline and post-treatment will be calculated.
Chronic Pain Self-Efficacy Score (CPSS) | CPSS will be assessed at baseline and at post-treatment, spanning approximately 4 months.
  Chronic Pain Self-Efficacy Score (CPSS) is a validated survey instrument that assesses an individual's beliefs and confident in their ability to manage and cope with chronic pain. Each item on the instrument is scored on a 10-point Likert Scale, from 10 (very uncertain) to 100 (very certain). Average subscale scores are calculated for each domain: self-efficacy for pain management (PSE), self-efficacy for coping with symptoms (CSE), and self-efficacy for physical function (FSE).

CONTACTS AND LOCATIONS:
Overall Officials: Jeungchan Lee, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Athinoula A. Martinos Center for Biomedical Imaging, Boston, Massachusetts, United States